CLINICAL TRIAL: NCT01120795
Title: Pegylated Interferon Alfa-2a Plus Ribavirin for Patients With Chronic Hepatitis c Virus on Opioid Pharmacotherapy: Virological and Psychological Outcomes
Brief Title: Pegylated Interferon and Ribavirin in Hepatitis C Patients on Opioid Pharmacotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: The University of New South Wales (Other); St Vincent's Hospital, Sydney (Other); Western Hospital, Australia (Other Government); Monash University (Other); Hoffmann-La Roche (Industry)
Responsible Party: Dr Joe Sasadeusz, Victorian Infectious Diseases Service, Royal Melbourne Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC 2000.175
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2010-05

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pegylated interferon and ribavirin (Experimental): Anti hepatitis C agents
  Interventions: Drug: Pegylated interferon and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon and ribavirin — Pegylated interferon 180 ug subcutaneous per week Ribavirin 1000-1200 mg /day for genotype 1 and 800 mg /day orally for genotype non 1 Duration: 48 weeks for genotype 1 and 24 weeks for gentoype non 1
  Other Names: Pegasys and Copegus
Drug: Pegylated interferon and ribavirin — Pegylated interferon 180 ug/ week subcutaneously Ribavrin 1000-1200 mg /day for genotype 1 and 800 mg/day orally for genotype 2 and 3 Treatment duration 48 weeks for genotype 1 and 24 weeks for genotypes 2 and 3
  Other Names: Pegasys and Copegus

SUMMARY:
The purpose of this study is to see if treatment of chronic hepatitis C in people who are on opiate replacement therapy such as methadone or buprenorphine (including patient who still inject drugs) is safe and effective.

DETAILED DESCRIPTION:
It is estimated that in excess of 170 million people worldwide are infected with the hepatitis C virus (HCV) resulting in 1.4 million deaths annually. In developed countries HCV is most commonly transmitted through injecting drug use (IDU) with estimates suggesting up to 80-90% of incident cases are due to unsafe injecting practices. Infection results in chronic infection in around 75% of cases and it is these patients who subsequently develop the life-threatening complications of liver failure and hepatocellular carcinoma due to progressive fibrosis.

Current standard of care consists of a combination of pegylated interferon and ribavirin which results in sustained virological response rates (SVR, defined as undetectable HCV RNA 24 weeks post treatment) in 54-63% of patients. This is strongly dependent on viral genotype with genotype 1 patients achieving lower SVR rates compared to genotype 2 and 3. These therapies are however associated with significant side effects, most notably psychiatric. Depression, anxiety and irritability are common and of concern is the attendant risk of suicidality in patients with a chronic illness in which depression is particularly common. Mood disorders have been reported to occur in up to 50% patients on therapy and can result in dose reductions and discontinuation in 40% and 20% patients respectively.

While more effective therapies have become available for the treatment of chronic HCV, they have not been largely utilised in patients actively injecting. This is due to concerns about potential poor adherence to treatment regimens, reinfection due to ongoing IDU, increased incidence of concomitant alcohol abuse, potential for increased side effects (especially psychiatric), concerns about pregnancy with ribavirin use due to non-adherence to contraception as well as active discrimination by practitioners. There are however considerable potential advantages including: improvement in the health of the infected individual, potential for decreasing the burden of disease to the community with its attendant costs as well as the potential for impact on transmission and its inherent potential public health benefits.

This multicentre study was conducted to determine the response rates as well as the AE profile and the psychiatric impact of therapy in a population with chronic hepatitis C (CHC) who were receiving opiate pharmacotherapy, many of who were still injecting.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. on opioid substitution therapy (methadone or buprenorphine)
3. serologic evidence of chronic hepatitis C infection determined by a detectable anti-HCV antibody for 6 months or greater with evidence of detectable HCV RNA
4. elevated ALT on at least two occasions at least one month apart within the past 6 months, with at least one during the screening period preceding the initiation of study drug dosing.
5. HCV treatment-naïve
6. Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection (unless contraindicated due to a bleeding disorder)
7. Compensated liver disease (Child-Pugh Grade A clinical classification).
8. All fertile males and females receiving ribavirin were required to be using two forms of effective contraception during treatment and during the 6 months after treatment
9. Women of child bearing potential were required to have a negative urine or blood pregnancy test documented within the 24-hour period prior to the first dose of study drug

Exclusion Criteria:

1. Women who were pregnant, breastfeeding or planning a pregnancy
2. Male partners of women who were pregnant
3. Patients who had previously received therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug
4. Recipients of any investigational drug 4 weeks or 5 half lives, whichever was longer, prior to the first dose of study drug
5. A positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, anti-HIV Ab
6. A history or other evidence of a medical condition associated with chronic liver disease other than HCV
7. Haemoglobin <12 g/dL in women or <13 g/dL in men, a neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening and serum creatinine level >1.5 times the upper limit of normal at screening.)
8. A history of a severe seizure disorder or current anticonvulsant use
9. Patients with a history of immunologically-mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, coronary artery disease, cerebrovascular disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
10. Patients with a history of thyroid disease which is poorly controlled on prescribed medications
11. Evidence of severe retinopathy
12. Evidence of excessive substance abuse as judged by the investigator
13. Patients with an increased baseline risk for anaemia (e.g. thalassaemia, spherocytosis, history of gastrointestinal bleeding, etc) or for whom anemia would be medically problematic.
14. Patients with a history of severe psychiatric disease (defined as acute phase of schizophrenia or bipolar disorder manic, mixed or depressive phase, severe anorexia, history of severe multiple episodes of self harm, currently screening as high or moderate suicide risk, current major depressive episode or current psychosis of any cause at screening)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-02; Primary Completion 2006-01 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks post cessation of HCV therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Sasadeusz, MBBS, Principal Investigator — Melbourne Health
Locations (4):
- Australia (4):
  - Nepean Hospital, Sydney, New South Wales
  - St Vincents Hospital, Sydney, New South Wales
  - Western Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Sasadeusz JJ, Dore G, Kronborg I, Barton D, Yoshihara M, Weltman M. Clinical experience with the treatment of hepatitis C infection in patients on opioid pharmacotherapy. Addiction. 2011 May;106(5):977-84. doi: 10.1111/j.1360-0443.2010.03347.x. PMID 21205057